CLINICAL TRIAL: NCT06194253
Title: Evaluation of the Reasons for Recourse and Diagnoses Associated With Early Recourse to an Emergency Structure After Initial Treatment Followed by a Return Home
Brief Title: Reasons for Recourse and Diagnoses Associated With Early Recourse to an Emergency Structure After Initial Treatment
Acronym: CallBack-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8958
Record Dates: First submitted 2023-12-15; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Urgent Care Centers
Keywords: Emergency Department; Urgent Care Centers
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To date, studies have been carried out on emergency department revisits but most are studies carried out in Anglo-Saxon territories. The studies carried out in France, for their part, concern the elderly geriatric population, or populations with specific pathologies such as child psychiatrists or patients with acute heart failure, but not the general adult population. Nevertheless, these studies have shown that knowledge of the risk factors for early readmission of a patient makes it possible to carry out targeted prevention actions in order to reduce this early recourse rate.

However, in a context of increasing emergency flow and increasing tension in the field with limited healthcare resources, returning home and outpatient care are increasingly favored. However, these strategies only make sense if outpatient follow-up is organized when early reconsultation is possible for certain indications that remain to be determined. In this context, it would be interesting to have information on the reasons for which patients return to the emergency room early after initial treatment. This would indeed make it possible to consider carrying out preventive actions in the long term in order to reduce this revisit rate on the one hand and on the other hand to identify the signs of seriousness which should bring the patient back to the emergency room as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Subject treated in the emergency room of the NHC or Hautepierre and having consulted the emergency room of one of the two sites 7 days after their first visit for an identical reason for recourse between January 1, 2017 to January 31, 2023.
* Patient who has not expressed his opposition to the reuse of his data for scientific research purposes.

Exclusion Criteria:

* Patient having expressed his opposition to the retrospective reuse of his data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - Major subject (≥18 years old) treated in the emergency room of the NHC or Hautepierre and having consulted the emergency room of one of the two sites 7 days after their first visit for an identical reason for recourse between January 1, 2017 to January 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of the most frequent reasons for recourse for which patients benefit from a new emergency consultation for the same reason within 7 days. | up to 7 days
  The aim of the study is to have information on the reasons for which patients return to the emergency room early after initial treatment. This would indeed make it possible to consider carrying out preventive actions in the long term in order to reduce this revisit rate on the one hand and on the other hand to identify the signs of seriousness which should bring the patient back to the emergency room as soon as possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Accueil des Urgences - CHU de Strasbourg - France, Strasbourg, France